CLINICAL TRIAL: NCT03532152
Title: Randomized, Prospective, Sham-controlled, Blinded, Cross-over Clinical Study of the Effect of the Virtual Reality (VR) Technology on Recovery of Indicators of the Autonomic Nervous System in Healthy Volunteers Affected by Moderate Stress
Brief Title: Study of the Effect of the VR Technology on Recovery of the Autonomic Nervous System in Volunteers Affected by Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pure Purr LLC (Other)
Collaborators: Pharmaxi LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PurePurr-001
Record Dates: First submitted 2018-05-02; First posted 2018-05-22 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Stress
Keywords: VR; moderate stress

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pure Purr VR technology (Active Comparator): The arm will use the virtual reality headset reproduces a dynamic video content that is visually perceived with the help of the high-resolution screen.
  The total length of the audio-video sequence is 6 minutes 11 seconds, of which 1 minute 11 seconds is the Pure Purr promotional video, and the duration of the investigational audio-visual sequence itself is 5 minutes.
  Interventions: Device: Pure Purr VR technology
- Sham VR technology (Sham Comparator): The arm will use the headset with audio-visual sequence is similar to the one in the investigational version of the software. The key difference is that the audio sequence has not been modified with the binaural effect and has not been synchronized with the tact of respiratory movements and the frequency of heart rate.
  The total length of the audio-video sequence is 6 minutes 11 seconds, of which 1 minute 11 seconds is the Pure Purr promotional video, and the duration of the investigational audio-visual sequence itself is 5 minutes.
  Interventions: Device: Sham VR technology

INTERVENTIONS:
Device: Pure Purr VR technology — The Pure Purr technology consists of BoboVR X1 headset with pre-installed software. The virtual reality headset reproduces a dynamic video content that is visually perceived with the help of the high-resolution screen. Also, the headset is able to play audio and transmit it via the headphones.
  The audio sequence has been modified by adding a binaural effect and has been synchronized with the tact of respiratory movements and the frequency of heart rate.
  Arms: Pure Purr VR technology
Device: Sham VR technology — The sham technology includes an identical BoboVR X1 virtual reality headset with pre-installed software. The audio-visual sequence is similar to the one in the investigational version of the software. The key difference is that the audio sequence has not been modified with the binaural effect and has not been synchronized with the tact of respiratory movements and the frequency of heart rate.
  Arms: Sham VR technology

SUMMARY:
The study assess the effect of the VR technology (Pure Purr technology) on the recovery of the autonomic nervous system in healthy volunteers affected by moderate stress. Study subject randomized into two groups: in Group 1 volunteers first be tested with the VR headset A, and during the next visit- headset B. Group 2 volunteers first be tested with the VR headset B, and during the next visit- headset A. Before, after and during VR session was conducted stress modulation and ECG recording.

The Pure Purr technology combines several audio and visual stimuli aimed at activation of the parasympathetic nervous system. Therefore, this study will investigate the effect of this technology on the recovery of autonomic nervous system performance after moderate stress.

DETAILED DESCRIPTION:
Pure Purr technology is based on discoveries in neurophysiology, medicine, acoustics, and computer engineering, which are used to initiate the physiological process of recreation, i.e. allostasis. Literally this term means "achieving stability through change". This is an active mechanism playing a part in normalization of the tone of the autonomic nervous system and maintaining stability of the body internal environment. The condition in which all our functions are implemented fully and sparingly in response to the load, and the level of adaptation remains high for a long time. Pure Purr is a software and hardware complex for relaxation and recreation based on a virtual reality headset with a display with sufficient resolution, built-in processor, memory, and extended-range stereo speakers. Positive effect on the cognitive function of the brain and the system of neurohumoral regulation is achieved due to the synchronous actuation of a number of stimuli, such as: visual sequence enhanced by the effect of virtual reality, harmonious music with the binaural rhythm technology, and modified cat purrs. Currently, the use of each technology is a scientifically proven trigger for the activation of individual parts of the human nervous system. And combining them in one software complex enhances the overall effect.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males 20-60 years old;
2. Volunteers have no history of cardiovascular diseases;
3. Volunteers have no essential abnormalities on the ECG;
4. Normal or moderate level of situational anxiety based on the Spielberger State-Trait Anxiety Inventory (STAI);
5. Signed Informed Consent Form for participation in the study.

Exclusion Criteria:

1. Intolerance to the VR technology;
2. HR 110 bpm or below 50 bpm;
3. RR above 23 breaths per minute;
4. Abuse of alcohol, psychotropic substances and narcotic agents;
5. Smoking more than 100 cigarettes a week;
6. Administration of medicinal products for the treatment of cardiovascular and nervous system diseases 3 days prior to participation in the study;
7. Drinking tonics and energy drinks for at least 2 hours prior to participation in the study;
8. Severe or acute forms of respiratory, urogenital, gastrointestinal, haematological, metabolic, endocrine, or neurological diseases;
9. Mental disorders, which, in the opinion of the investigator, may distort the results of the study;
10. Participation in any clinical study over the last 3 months prior to enrolment to the study;
11. Parkinson's disease, Parkinson's symptoms, tremor, restless leg syndrome, and other motility disorders;
12. Pregnancy;
13. Any disease of the thyroid gland.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Power in high frequency range (HF) [ms2] | The outcome measure will be assessed between two visits with minimum interval 24 up to seven days
  Change from Power in high frequency range (HF) [ms2] at 5 minutes before and after VR technology using

SECONDARY OUTCOMES:
The square root of the mean of the sum of the squares of differences between adjacent NN intervals (rMSSD), [ms] | The outcome measure will be assessed between two visits with minimum interval 24 up to seven days
  Change from rMSSD variable at 5 minutes before and after VR technology using
Standard deviation of all NN intervals (SDNN), [ms] | The outcome measure will be assessed between two visits with minimum interval 24 up to seven days
  Change from SDNN variable at 5 minutes before and after VR technology using
Ratio Power in low frequency range [ms2]/ Power in high frequency range [ms2] (Ratio LF [ms2]/HF [ms2]) | The outcome measure will be assessed between two visits with minimum interval 24 up to seven days
  Change from Ratio LF [ms2]/HF [ms2] at 5 minutes before and after VR technology using
Total power (TP), [ms2] | The outcome measure will be assessed between two visits with minimum interval 24 up to seven days
  Change from Total power (TP) variable at 5 minutes before and after VR technology using
Heart Rate (HR) variable. | The outcome measure will be assessed between two visits with minimum interval 24 up to seven days
  Change from Heart Rate (HR) variable at 5 minutes before and after VR technology using
BP (both systolic and diastolic blood pressure) variable. | The outcome measure will be assessed between two visits with minimum interval 24 up to seven days
  Change from systolic and diastolic blood pressure at 5 minutes before and after VR technology using
Spielberger state-trait anxiety inventory (STAI) variable. | The outcome measure will be assessed between two visits with minimum interval 24 up to seven days
  Change from STAI variable at 5 minutes before and after VR technology using. STAI-Examination of the level of situational anxiety.
  Statement for еxamination:
  1. Calm down
  2. Safe
  3. Tense
  4. Annoyed
  5. Comfortable
  6. Upset
  7. Concerned with future misfortunes
  8. Relaxed
  9. Anguished
  10. At ease
  11. Self-confidence
  12. Nervous
  13. Restless
  14. Downhearted
  15. Rested
  16. Satisfied
  17. Concerned
  18. Stunned
  19. Happy
  20. I fell good
  The range for each subscale from 1 to 4 point.
  Processing of results:
  Calculate the total score based on answers given by volunteers.
  While interpreting the results, use the following levels of anxiety:
  * up to 30 points - low,
  * 31 - 44 points - moderate;
  * 45 and more - high.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Aganov, Ph.D., Principal Investigator — Dr. Sam LLC
Locations (1):
- Doctor Sam Medical Network, Kyiv, Kyiv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT03532152/Prot_000.pdf